CLINICAL TRIAL: NCT00537784
Title: Platelet Concentrate in Achilles Tendon Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Per Aspenberg, professor, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Trombocytakilles
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Achilles Tendon Rupture; Soft Tissue Injury; Tendon Injury
Keywords: platelets tendon ligament
MeSH Terms: conditions — Soft Tissue Injuries; Tendon Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Injection of autologous platelet concentrate into repair site
  Interventions: Biological: Autologous platelets
- 2 (Placebo Comparator): No injection
  Interventions: Biological: no injection

INTERVENTIONS:
Biological: Autologous platelets — Local injection 10mL, about 2.5 x 10E10 platelets.
  Arms: 1
Biological: no injection
  Arms: 2

SUMMARY:
People operated for a rupture of the Achilles tendon receive a concentrate of their own platelets injected into the operated area. The study is randomized and single-blinded, with 20 treated patients and 20 controls, who get no injection. The primary endpoint is a mechanical property of the tendon after 12 weeks (modulus of elasticity), as measured by a special type of radiography. This radiography uses 0.8 mm metal markers, which are injected into the tendon. The tendon is mechanically loaded during radiography and its strain can be measured as increased distance between the markers. Other mechanical variables at 6, 12 and 52 weeks are secondary variables, as well as a validated patient-administrated questionaire at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Achilles tendon rupture, age 18-65.

Exclusion Criteria:

* Any counterindication for surgical treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Modulus of elasticity | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: per aspenberg, Principal Investigator — University of Linköping
Locations (1):
- Univ Hosp, Linköping, Sweden

REFERENCES:
- [Result] Schepull T, Kvist J, Norrman H, Trinks M, Berlin G, Aspenberg P. Autologous platelets have no effect on the healing of human achilles tendon ruptures: a randomized single-blind study. Am J Sports Med. 2011 Jan;39(1):38-47. doi: 10.1177/0363546510383515. Epub 2010 Nov 3. PMID 21051425